CLINICAL TRIAL: NCT02973243
Title: The Vital Signs to Identify, Target, and Assess Level (VITAL) Care Study III
Status: Completed | Type: Observational
Sponsor: Philips Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: YGB-816-VITALIII
Record Dates: First submitted 2016-11-22; First posted 2016-11-25 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Cardiac Arrest; Renal Failure; Respiration Failure; Myocardial Infarction; Severe Sepsis
Keywords: early warning scoring; respiration rate; acute care teams; NEWS; CREWS
MeSH Terms: conditions — Heart Arrest; Renal Insufficiency; Respiratory Insufficiency; Myocardial Infarction; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Manual Respiration Rate Measurement: Patients with manually measured respiratory rate
- Automatic Respiration Rate Measurement: Patients with automatically measured respiratory rate
  Interventions: Device: Automatic RR Measurement

INTERVENTIONS:
Device: Automatic RR Measurement — Different newly developed respiration rate sensors are applied at the bedside during the intervention phase which send data to the IntelliVue Guardian System.
  Groups: Automatic Respiration Rate Measurement

SUMMARY:
To evaluate the effect of automated recording on frequency of recorded scores, number of automated notifications and serious events.

DETAILED DESCRIPTION:
The frequency of EWS scores, number of automated notifications and serious events performed on a general ward is contingent on the quality and frequency of vital signs measurement like respiratory rate. This is due to the EWS escalation schemes of hospitals with an acute intervention team. Obtained sub-score trigger levels of vital signs contribute to higher and more frequent scoring.

We examine the influence of different respiration rate sensor concepts and measurements on scoring (NEWS and CREWS) and workflow in a typical UK gastroenterology and respiratory ward.

ELIGIBILITY:
Inclusion Criteria:

* patients admitted to the study units during the period of data collection

Exclusion Criteria:

* palliative patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators plan to observe a non-probability, convenience sample of patients which will consist primarily of acutely ill hospitalized adult patients (at least 18 years of age). Study participants will be recruited from all eligible patients during the enrollment period who are having vital signs monitoring performed as Standard of Care.
Sampling Method: Non-Probability Sample
Enrollment: 446 (Actual)
Dates: Start 2016-10-05 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
Number of NEWS Scores | 8-12 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Christian P Subbe, MD, Principal Investigator — Ysbyty Gwynedd Hospital
Locations (1):
- Ysbyty Gwynedd Hospital, Bangor, United Kingdom

IPD SHARING:
Plan to Share IPD: No